CLINICAL TRIAL: NCT03181373
Title: Longitudinal Descriptive Study of the Correlation Between Cognitive Functions, White Matter Anatomical Pathways and Functional Magnetic Resonance Imaging Activations in Patients With Moderate to Severe Head Trauma.
Brief Title: IRM Cognition in Patients With Head Trauma
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Clementel (Unknown); Maurice Gantchoula (Unknown); LADAPT (Other); APF (Unknown)
Responsible Party: Sponsor
Other Study IDs: CHU-328
Record Dates: First submitted 2017-05-09; First posted 2017-06-08 (Actual); Last update posted 2017-06-08 (Actual); Status verified 2017-05

CONDITIONS: Brain-damaged Patients
Keywords: Craniocerebral injury; Mild and severe brain traumatic injury; Neuropsychological abilities; Clinical assessment; Anatomical and functional imaging
MeSH Terms: conditions — Craniocerebral Trauma; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Traumatic brain injury population: Defined population : traumatic brain injury population
  Interventions: Other: Cognitive rehabilitation program

INTERVENTIONS:
Other: Cognitive rehabilitation program — Rehabilitation

SUMMARY:
Longitudinal descriptive study of a cohort of twenty brain-damaged patients for a two years period.

DETAILED DESCRIPTION:
The following data are collected in 3 months, 12 months then 24 months after the accident with followed data collection :

* Clinical, neuropsychological assessments
* Diffusion magnetic resonance imaging (MRI) for the reconstruction of anatomical pathways
* Functional imaging data.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, over the age of 18.
* Mild traumatic brain injury (Initial Glasgow score between 9 and 12)
* Severe brain injury (Initial Glasgow score between 3 and 8),
* Diffuse axonal injury and/or focal lesions.

Exclusion Criteria:

* Patients with MRI contraindications,
* Antecedents of brain lesions,
* Important lesions of the lobes and cortex on cerebral CT,
* Anoxic lesions related to cardiorespiratory arrest,
* Must be able to perform neuropsychological tests,
* Visual and auditory impairments.
* Aphasia

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with traumatic brain injury
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2014-09-26 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Baseline standardized volume of the white matter fascicles | at 3, 12 and 24 months
  determined on the "iplan" software. Baseline measured at 3 months after brain traumatic injury.

SECONDARY OUTCOMES:
Measure of the volume of activations clusters | at 3, 12 and 24 months
  during functional MRI for attention, motor, working memory, language tasks.
Location of activation clusters | at 3, 12 and 24 months
  during functional MRI for attention, motor, working memory, language tasks.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, Auvergne, France